CLINICAL TRIAL: NCT00313404
Title: Assessment of Calicivirus Survival in Surface Water and Subsurface Water
Brief Title: Infectivity of Norovirus in Groundwater-Human Challenge Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Christine Moe, PhD, Gangarosa Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 0584-2002; EPA-5 R01 AI056351-03 (Other: Emory University Clinical Trials Office); 82911601-1 (Other Grant/Funding Number: Environmental Protection Agency); RSPHGH-CLM-2005-EPANoV (Other: Other)
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Norovirus; Gastroenteritis; Clinical Trial; Stomach flu
MeSH Terms: conditions — Gastroenteritis | interventions — Groundwater

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norovirus in groundwater (Experimental): We dosed volunteers with safety tested infectious norovirus in groundwater (that met EPA standards for drinking water). The length of time norovirus remained in groundwater varied by volunteer.
  Interventions: Biological: Safety tested norovirus inoculum

INTERVENTIONS:
Biological: Safety tested norovirus inoculum — This is a safety tested live infectious norovirus inoculum that has been placed in groundwater that meets EPA drinking water standards
  Other Names: Norwalk virus in groundwater

SUMMARY:
Norwalk virus and related "Norwalk-like viruses" are the most common cause of outbreaks of stomach sickness (nausea, vomiting, diarrhea) in older children and adults in the United States. These viruses are sometimes found in drinking water, ice, shellfish and in other foods. They can be spread easily from contact with water, food, objects or hands that have even small amounts of feces from someone who was sick.

The purpose of this research study is to see how long Norwalk virus can survive in water and still be able to cause sickness. When this is determined the researchers will be able to recommend risk levels for norovirus contaminated waters. Another purpose for this study is to see how a person's body's immune cells respond to Norwalk virus in the body. During this study volunteers will receive a dose of Norwalk virus in water that may make them sick.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Must be within 33% of normal body mass index

Exclusion Criteria:

* Have a job in which they handle food
* Work in a child care, elderly care center or if they live with young children or anyone who has a weak immune system
* Are not willing or able to wash their hands every time after they go to the bathroom, or before and after they prepare or handle food for up to eight days after they take the virus
* Are over the age of 50
* Are pregnant
* Have tested positive for the HIV virus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Infection with norovirus | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Christine Moe, PhD, Principal Investigator — Emory University; George M Lyon III, MD, MMSc, Principal Investigator — Emory University; Kellogg Schwab, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Emory University General Clinical Research Center, Atlanta, Georgia, United States

REFERENCES:
- [Result] Seitz SR, Leon JS, Schwab KJ, Lyon GM, Dowd M, McDaniels M, Abdulhafid G, Fernandez ML, Lindesmith LC, Baric RS, Moe CL. Norovirus infectivity in humans and persistence in water. Appl Environ Microbiol. 2011 Oct;77(19):6884-8. doi: 10.1128/AEM.05806-11. Epub 2011 Aug 19. PMID 21856841
- [Derived] Williams AM, Ladva CN, Leon JS, Lopman BA, Tangpricha V, Whitehead RD, Armitage AE, Wray K, Morovat A, Pasricha SR, Thurnham D, Tanumihardjo SA, Shahab-Ferdows S, Allen L, Flores-Ayala RC, Suchdev PS. Changes in micronutrient and inflammation serum biomarker concentrations after a norovirus human challenge. Am J Clin Nutr. 2019 Dec 1;110(6):1456-1464. doi: 10.1093/ajcn/nqz201. PMID 31504095